CLINICAL TRIAL: NCT00534664
Title: Phase II Study to Determine the Effectiveness of Intrabuccally Administered Amplitude-Modulated Electromagnetic Fields in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Phase I/II Study of Amplitude-Modulated Electromagnetic Fields in the Treatment of Advanced Hepatocellular Carcinoma
Acronym: TheraBionic
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THBC-HCC-01
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TheraBionic device — Daily outpatient treatment with theraBionic device

SUMMARY:
The goal of this study is to investigate the safety and feasibility of treating patients with advanced hepatocellular carcinoma with a noninvasive device administering low level of amplitude-modulated electromagnetic fields.

ELIGIBILITY:
Inclusion Criteria:

* Advanced biopsy-proven HCC
* Performance status ECOG 0-1
* Patients with Child Pugh A and B cirrhosis scores
* Absence of medical or psychiatric contraindication which, in the opinion of the treating investigator, would make the patient's participation in this trial inappropriate.
* Presence of one or more measurable lesion(s) according to the RECIST criteria.
* Lesions treated with chemoembolization or ablation by means of radio frequencies will not be considered measurable in this study.
* Patients on a liver transplant waiting list may be included
* Patient must not have curative treatment options other than liver transplant
* Patient may have been treated with intrahepatic treatment (chemoembolization or intrahepatic chemotherapy) or conventional chemotherapy or sorafenib or other experimental therapies prior to study entry. There is no limit for the number of prior therapies
* Extra hepatic metastases do not constitute an exclusion criterion, except for active CNS metastases.
* At least 4 weeks must have elapsed since administration of any anti-cancer treatment.
* Other anti-cancer treatments are not permitted during this study
* Patients must be more than 18 old and must be able to understand and sign an informed consent.
* Patient must agree to be followed up according to the study protocol.
* Patients may have either stable disease or disease progression according to the principal investigator assessment.
* Patients who carry a pacemaker or any other implantable electronic device are not allowed in the study

Exclusion Criteria:

* Suspected or biopsy confirmed brain metastases
* Patients with hepatic cirrhosis with Child-Pugh class C
* Patients who have received a liver transplant.
* Patients who had a surgical resection of the disease and who do not have measurable disease.
* Pregnant women
* Patients who still show objective response (complete or partial response) according to the RECIST criteria due to the last anti-cancer therapy
* Patients diagnosed with another type of cancer (excluding basal cell carcinoma) during the last five last years or whose cancer diagnosed previously is not in remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederico P Costa, MD, Principal Investigator — Disciplina de Transplante e Cirurgia do Fígado
Locations (1):
- Disciplina de Transplante e Cirurgia do Fígado, São Paulo, São Paulo, Brazil